CLINICAL TRIAL: NCT06325267
Title: A Single Center, Retrospective Clinical Study on the Clinical Characteristics of Primary Liver Cancer
Brief Title: Clinical Characteristics of Primary Liver Cancer
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jie Li, Principal investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: PLC
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Primary Liver Cancer
Keywords: primary liver cancer; clinical features
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary liver cancer (PLC) is the sixth most common malignancy in the world and the third most common cause of malignancy death. In 2020, there were about 905,677 new cases of PLC worldwide, and 830,180 deaths. Despite the availability of a variety of treatments for PLC, the 5-year net survival rate is still only 5% to 30%. How to effectively reduce the disease burden of PLC is a major public health problem that needs to be solved worldwide. The clinical characteristics and prognosis of PLC caused by different pathogenic factors are different. Therefore, it is of great significance to fully identify the risk factors of PLC, be familiar with the clinical characteristics and prognosis of disease development, and understand the relevant monitoring and follow-up strategies for the prevention and treatment of PLC.

DETAILED DESCRIPTION:
Primary liver cancer (PLC) is the sixth most common malignancy in the world and the third most common cause of malignancy death. PLC mainly includes hepatocellular carcinoma (75%-85%) and intrahepatic cholangiocarcinoma (10%-15%). In 2020, there were about 905,677 new cases of PLC worldwide, and 830,180 deaths. Despite the availability of a variety of treatments for PLC, the 5-year net survival rate is still only 5% to 30%. How to effectively reduce the disease burden of PLC is a major public health problem that needs to be solved worldwide. Common risk factors for PLC include Hepatitis B virus (HBV), Hepatitis C virus (HCV) infection, alcohol consumption, metabolic factors, etc. Although antiviral drugs can control or even cure chronic HBV and HCV to a certain extent, chronic viral infection is still the leading cause of PLC worldwide. In addition, with the prevalence of obesity, diabetes and non-alcoholic fatty liver disease (NAFLD), the incidence of non-infectious PLC is gradually increasing. In recent years, NAFLD has gradually become the leading cause of liver transplant waiting list for patients with hepatocellular carcinoma in the United States. The clinical characteristics and prognosis of PLC caused by different pathogenic factors are different. Therefore, it is of great significance to fully identify the risk factors of PLC, be familiar with the clinical characteristics and prognosis of disease development, and understand the relevant monitoring and follow-up strategies for the prevention and treatment of PLC. Currently, there are few large, single-center cohort studies on the clinical features and long-term prognosis of PLC.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older;
2. initial diagnosis of primary liver cancer based on enhanced CT or enhanced MRI or pathology

Exclusion Criteria:

1. other types of malignant tumors;
2. mental illness, severe cardiopulmonary dysfunction, severe renal insufficiency, serious infection and cerebrovascular accident;
3. received liver transplant or other organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary liver cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Epidemiological characteristics of overall cohort by liver disease etiology | 0 year
  Epidemiological characteristics of overall cohort by liver disease etiology, including HBV, HCV, NAFLD, ALD and others.
Clinical characteristics of overall cohort by liver disease etiology | 0 year
  Clinical characteristics of overall cohort by liver disease etiology, including HBV, HCV, NAFLD, ALD and others.

SECONDARY OUTCOMES:
Survival rates of overall cohort and different etiologies | 1 year, 3years，10 years
  1-year, 3-year, 5-year, and 10-year survival rates for overall cohort and different etiologies
Risk factors of prognosis in overall cohort and different etiologies | 10 years
  Risk factors for recurrence, metastasis, and all cause death in overall cohort and different etiologies

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China